CLINICAL TRIAL: NCT03691324
Title: Could Training in Inhalation Technique During the Hospital Stay and Discharge Services From the Pharmacy Reduce the Rate of Readmissions for COPD Patients? - A Pilot Study
Brief Title: Training of Inhalation Technique in Hospitalized Chronic Obstructive Pulmonary Disease (COPD) Patients - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University College (Other)
Collaborators: Oslo University Hospital (Other); Hospital Pharmacy Enterprise, South Eastern Norway (Other)
Responsible Party: Principal Investigator, Liv Mathiesen, Associate professor, Oslo University College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2018/753
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients receive an inhalation technique education based on standardized procedure developed by The Norwegian Pharmacy Association. In addition they are offered a discharge service day before or the day of discharge; a second inhalation training and dispensing of their prescribed COPD- medicines.
  Interventions: Other: Inhalation technique training and discharge service
- Standard care (No Intervention): Patients receive standard care and follow up of their COPD-treatment

INTERVENTIONS:
Other: Inhalation technique training and discharge service — Patient drug counselling one-to-one, focusing on inhalation drugs and technique
  Arms: Intervention

SUMMARY:
Inhalation drugs are essential in the treatment of COPD, in controlling symptoms and preventing exacerbations. The aim of this pilot study is to collect data necessary for the planning of future efficacy trials. We plan to assess the value of providing training in inhalation technique to hospitalized COPD patients. Data on rehospitalizations will be collected from the hospital's medical records and from the National Patient Registry . The inhalation technique of all recruited patients will de assessed at baseline. The patients will then be randomised 1:1 to the intervention or standard care group. The intervention consists of a drug counselling, focusing on inhalation technique. In addition patients in the intervention group will have their medicines personally delivered from the hospital pharmacy at discharge (discharge service). Patients will be asked to fill in questionnaires evaluating the inhalation training and the discharge service

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the pulmonary ward, the Medical Department, Oslo University Hospital, Oslo, Norway

Exclusion Criteria:

Patients

* previously included to the study
* usually not administering their inhalation drugs themselves
* using nebulizer chamber with their drug
* who are contagious, thus restricting accessibility of personnel
* who are not able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Time to first readmission | One year after discharge of the last patient
  Time to readmission based on data from the national patient registry

SECONDARY OUTCOMES:
Improvement in patient reported symptom score (CAT-score) from baseline to 2 months after discharge | 2 months after discharge
  COPD assessment test (CAT) scores at baseline and 2 months after discharge.
Proportion of patients readmitted 3 months after discharge | 3 months
  Based on the hospital records. Preliminary data to be published in a master thesis, as the data on the primary endpoint will be received too late

CONTACTS AND LOCATIONS:
Overall Officials: Liv Mathiesen, PhD, Principal Investigator — Oslo University Collage
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Sharing of individual patient data is not allowed by the approving authority

REFERENCES:
- [Derived] Kebede AT, Trapnes E, Lea M, Abrahamsen B, Mathiesen L. Effect of pharmacist-led inhaler technique assessment service on readmissions in hospitalized COPD patients: a randomized, controlled pilot study. BMC Pulm Med. 2022 May 27;22(1):210. doi: 10.1186/s12890-022-02004-z. PMID 35624509